CLINICAL TRIAL: NCT03814031
Title: Hepatic Vein Flow Assessment With Transesophageal Echocardiography for Postoperative Graft Function Prediction in Orthotopic Liver Transplantation
Brief Title: Hepatic Vein Flow During Orthotopic Liver Transplantation as Predictive Factor for Postoperative Graft Function
Status: Completed | Type: Observational
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Yoshihisa Morita, MD, Henry Ford Health System
Other Study IDs: 12156
Record Dates: First submitted 2019-01-16; First posted 2019-01-23 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-05

CONDITIONS: Postoperative Graft Function
Keywords: TEE; orthotopic liver transplant; EAD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EAD after orthotopic liver transplantation: Early allograft dysfunction (EAD), which was defined by the presence of one or more of the following: total bilirubin (t-bil) ≥ 10 mg/dL (171 μmol/L) or, INR ≥ 1.6 on day 7, and ALT/AST > 2,000 IU/L within the first 7 days.
  Interventions: Other: NO internvention
- No EAD after orthotopic liver transplantation: No EAD
  Interventions: Other: NO internvention

INTERVENTIONS:
Other: NO internvention — NO internvention

SUMMARY:
Hepatic vein flow (HVF) assessment using transesophageal echocardiography (TEE) has a potential to predict postoperative graft function in orthotopic liver transplant (OLT). Investigators will measure HVF using TEE and assess the correlation with postoperative graft function indices such as early allograft dysfunction(EAD), prolonged INR, platelet, and total bilirubin.

DETAILED DESCRIPTION:
During OLT, intraoperative TEE assessment of HVF (systolic and diastolic) were measured, and adjusted with donor graft weight. This index, HVF index, was assessed for correlation with EAD. HVF was calculated with hepatic vein area (cm2) x hepatic vein velocity (ml/s) in systole and diastole during the neohepatic phase. Investigators did ROC analysis to assess the predictive power for EAD, prolonged INR, platelet, and total bilirubin.

ELIGIBILITY:
Inclusion Criteria:

Orthotopic liver transplants which uses TEE intraoperatively Must be Piggy back technique

-

Exclusion Criteria:

TEE absolute contraindication patient refusal

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: OLT with piggy back technique
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoshihisa Morita, MD, Principal Investigator — Henry Ford Hospital
Locations (1):
- HFHS, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- EAD After Orthotopic Liver Transplantation: Early allograft dysfunction (EAD), which was defined by the presence of one or more of the following: total bilirubin (t-bil) ≥ 10 mg/dL (171 μmol/L) or, INR ≥ 1.6 on day 7, and ALT/AST > 2,000 IU/L within the first 7 days.
  NO intervention
- No EAD After Orthotopic Liver Transplantation: No EAD noted after orthotopic liver transplantation
  NO intervention
Period: Overall Study
Arm/Group | EAD After Orthotopic Liver Transplantation | No EAD After Orthotopic Liver Transplantation
Started | 26 | 71
Completed | 26 | 71
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Of 120 potentially eligible patients, 97 patients participated in the study (patient refusal to participate in the study: 2 cases, absolute TEE contraindication: 5 cases, damping of the HVs images: 6 cases, and technically challenging to obtain appropriate views for HVF measurement: 10 cases).
Groups:
- Total: Total of all reporting groups
Arm/Group | EAD After Orthotopic Liver Transplantation | No EAD After Orthotopic Liver Transplantation | Total
Number analyzed (Participants) | 26 | 71 | 97
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 41 | 51
  >=65 years | 16 | 30 | 46
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 58 [45 to 64.5] | 55 [50.8 to 64] | 56 [47 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 28 | 39
  Male | 15 | 43 | 58
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 26 | 71 | 97

OUTCOME MEASURES:

1. Primary Outcome: EAD
Description: Primary outcome was early allograft dysfunction (EAD), which was defined by the presence of one or more of the following: total bilirubin (t-bil) ≥ 10 mg/dL (171 μmol/L) or, INR ≥ 1.6 on postoperative day 7. and ALT/AST > 2,000 IU/L
  Systolic and diastolic hepatic vein flow index was assessed intraoperatively in neohepatic phase in both of EAD and non EAD group, and reported.
Time Frame: EAD met at any point within the first 7 days status post OLT
Measure: Median (Inter-Quartile Range); unit: L/kg/min
Arm/Group | EAD After Orthotopic Liver Transplantation | No EAD After Orthotopic Liver Transplantation
Number analyzed (Participants) | 26 | 71
L/kg/min
  HV flow systolic index | 1.23 [0.85 to 1.73] | 2.19 [1.28 to 3.7]
  HV flow diastolic index | 0.87 [0.62 to 1.32] | 1.54 [1.07 to 2.34]

2. Secondary Outcome: Acute Rejection
Description: Acute rejection noted with biopsy at any point within 6 to 8 weeks post-transplant
Time Frame: Acute rejection noted at any point within 6-8 weeks post transplant
Population: Adult patients undergoing the orthotopic liver transplant piggy-back technique with TEE-measured HV flow
Measure: Median (Inter-Quartile Range); unit: L/kg/min
Groups:
- Acute Rejrection: Acute rejection noted with biopsy within 6 to 8 weeks post-transplant
- No Acute Rejection: NO sign of acute rejection or acute rejection noted with biopsy within 6 to 8 weeks post-transplant
Arm/Group | Acute Rejrection | No Acute Rejection
Number analyzed (Participants) | 8 | 5
L/kg/min
  HV flow systolic index | 0.738 [0.690 to 1.341] | 1.535 [0.844 to 2.570]
  HV flow diastolic index | 0.571 [0.570 to 1.024] | 1.101 [0.708 to 1.644]

3. Secondary Outcome: Prolonged (>Seven Days) Time to Normalize Total Bilirubin (TIME T-bil)
Description: Normal total bilirubin < 1.2 mg/dL
Time Frame: postoperative day 7 assessment
Population: Adult patients undergoing the orthotopic liver transplant piggy-back technique with TEE-measured HV flow
Measure: Median (Inter-Quartile Range); unit: L/kg/min
Groups:
- Prolonged (>Seven Days) Time to Normalize Total Bilirubin (TIME T-bil): Normal total bilirubin < 1.2mg/dL
- No Prolonged (>Seven Days) Time to Normalize Total Bilirubin (TIME T-bil): Time to normalize total bilirubin < 7 days
  Normal total bilirubin < 1.2 mg/dL
Arm/Group | Prolonged (>Seven Days) Time to Normalize Total Bilirubin (TIME T-bil) | No Prolonged (>Seven Days) Time to Normalize Total Bilirubin (TIME T-bil)
Number analyzed (Participants) | 52 | 45
L/kg/min
  HV flow systolic index | 1.086 [0.691 to 1.438] | 2.051 [1.077 to 2.868]
  HV flow diastolic index | 0.806 [0.469 to 1.040] | 1.351 [0.954 to 2.186]

4. Secondary Outcome: Prolonged (>Seven Days) Time to Normalize INR (TIME Inr)
Description: Normal INR < 1.16
Time Frame: postoperative day 7 assessment
Population: Adult patients undergoing the orthotopic liver transplant piggy-back technique with TEE-measured HV flow
Measure: Median (Inter-Quartile Range); unit: L/kg/min
Groups:
- Prolonged (>Seven Days) Time to Normalize INR (TIME Inr): Nornal INR < 1.16
- No Prolonged (>Seven Days) Time to Normalize INR (TIME Inr): Time to normalize INR (TIME inr) < 7days
  NOrmal INR < 1.16
Arm/Group | Prolonged (>Seven Days) Time to Normalize INR (TIME Inr) | No Prolonged (>Seven Days) Time to Normalize INR (TIME Inr)
Number analyzed (Participants) | 35 | 62
L/kg/min
  HV flow systolic index | 1.081 [0.639 to 1.604] | 1.484 [0.736 to 2.518]
  HV flow diastolic index | 0.954 [0.526 to 1.222] | 1.050 [0.666 to 1.526]

5. Secondary Outcome: Prolonged (>Seven Days) Time to Normalize Platelet Count (TIME Plt).
Description: Normal platelet count > 140 B/L
Time Frame: postoperative day 7 assessment
Population: Adult patients undergoing the orthotopic liver transplant piggy-back technique with TEE-measured HV flow
Measure: Median (Inter-Quartile Range); unit: L/kg/min
Groups:
- Prolonged (>Seven Days) Time to Normalize Platelet Count (TIME Plt)): Normal platelet count > 140 B/L
- No Prolonged (>Seven Days) Time to Normalize Platelet Count (TIME Plt): Time to normalize platelet count< 7 days
  Normal platelet count > 140 B/L
Arm/Group | Prolonged (>Seven Days) Time to Normalize Platelet Count (TIME Plt)) | No Prolonged (>Seven Days) Time to Normalize Platelet Count (TIME Plt)
Number analyzed (Participants) | 75 | 22
L/kg/min
  HV flow systolic index | 1.341 [0.690 to 2.243] | 1.379 [0.867 to 2.553]
  HV flow diastolic index | 0.829 [0.713 to 1.98] | 1.024 [0.580 to 1.470]

6. Post Hoc Outcome: Intra-rater Reliability Analyses of HVFi
Description: Intra-rater and inter-rater reliability analyses of HVFi are performed using intraclass correlation coefficient (ICC). We randomly pick up 30 images and obtain consistency ICC for inter-observer variability using all three investigators (A, B, and C), and absolute-agreement ICC for intra-observer variability using investigator C, who measure all images twice with an interval between 6 and 8 weeks.
  For inter-observer variability, 3 investigators post-hoc determine HVFi based on the pulse-wave Doppler signal.
Time Frame: Timing is postoperatively at any point 6-8 weeks. Duration is a day.
Population: Randomly chosen 30 patients among enrolled patients
Measure: Median (95% Confidence Interval); unit: ICC
Groups:
- HVFi Systolic; HVFi Diastolic: We calculate HVF as follows: HVF (L/min) = HV area (cm2) x HV max velocity (cm/s) in systole and diastole x 60/1000, where HV area (cm2) = square of HV radius (cm) x 3.14, and HV max velocity (cm/s) is measured by TEE PWD with sample volume selected in the HV, where diameter of HV is measured as well. Efforts are made to align PWD and HV. We define HV flow index (HVFi) as HVF/donor liver weight (kg).
Arm/Group | HVFi Systolic | HVFi Diastolic
Number analyzed (Participants) | 30 | 30
ICC | 0.998 [0.997 to 0.999] | 0.998 [0.996 to 0.999]

7. Post Hoc Outcome: Inter-rater Reliability Analyses of HVFi
Description: Intra-rater and inter-rater reliability analyses of HVFi are performed using intraclass correlation coefficient (ICC). We randomly pick up 30 images and obtain consistency ICC for inter-observer variability using all three investigators (A, B, and C). For inter-observer variability, 3 investigators post-hoc determine HVFi based on the pulse-wave Doppler signal.
Time Frame: Timing is postoperative at any point. Duration is a day.
Population: Randomly chosen 30 patients among enrolled patients
Measure: Mean (95% Confidence Interval); unit: ICC
Arm/Group | HVFi Systolic | HVFi Diastolic
Number analyzed (Participants) | 30 | 30
ICC | 0.997 [0.995 to 0.998] | 0.993 [0.988 to 0.996]

ADVERSE EVENTS:
Time Frame: 3 months postoperatively
Description: No research related adverse events occurred. Since this is additional measurement of hepatic vein flow using existing TEE, no adverse events were anticipated or occurred.
Groups:
- EAD After Orthotopic Liver Transplantation: Early allograft dysfunction (EAD), which was defined by the presence of one or more of the following: total bilirubin (t-bil) ≥ 10 mg/dL (171 μmol/L) or, INR ≥ 1.6 on day 7, and ALT/AST > 2,000 IU/L within the first 7 days.
  NO internvention
- No EAD After Orthotopic Liver Transplantation: No EAD group.
  NO intervention
Arm/Group | EAD After Orthotopic Liver Transplantation | No EAD After Orthotopic Liver Transplantation
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/76
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/71
Other Adverse Events (participants affected / at risk) | 0/26 | 0/71

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-18): https://cdn.clinicaltrials.gov/large-docs/31/NCT03814031/Prot_SAP_000.pdf
  • Informed Consent Form (2019-03-18): https://cdn.clinicaltrials.gov/large-docs/31/NCT03814031/ICF_001.pdf